CLINICAL TRIAL: NCT02570165
Title: Study 201012: A Dose-Finding Study of Batefenterol (GSK961081) Via Dry Powder Inhaler in Patients With COPD
Brief Title: Dose-Finding Study of Batefenterol (GSK961081) Via Dry Powder Inhaler in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201012; 2015-001409-15 (EudraCT Number)
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: efficacy; dry powder inhaler; vilanterol; batefenterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol; GSK573719; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Batefenterol 37.5 mcg (Experimental): Each subject will receive batefenterol 37.5 mcg (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Batefenterol
- Batefenterol 75 mcg (Experimental): Each subject will receive batefenterol 75 mcg (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Batefenterol
- Batefenterol 150 mcg (Experimental): Each subject will receive batefenterol 150 mcg (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Batefenterol
- Batefenterol 300 mcg (Experimental): Each subject will receive batefenterol 300 mcg (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Batefenterol
- Batefenterol 600 mcg (Experimental): Each subject will receive batefenterol 600 mcg (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Batefenterol
- UMEC/VI 62.5/25 mcg (Experimental): Each subject will receive UMEC/VI 62.5/25 mcg (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Umeclidinium/ Vilanterol
- Placebo (Experimental): Each subject will receive placebo (1 actuation) once daily via DPI in the morning for 42 days of treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Batefenterol — Batefenterol will be provided as dry white powder for inhalation via a DPI with 30 doses (2 strips with 30 blisters per strip). First strip will contain lactose and the second strip will contain batefenterol blended with lactose with a unit dose strength of 37.5 mcg, 75 mcg, 150 mcg, 300 mcg, or 600 mcg per blister
  Arms: Batefenterol 150 mcg; Batefenterol 300 mcg; Batefenterol 37.5 mcg; Batefenterol 600 mcg; Batefenterol 75 mcg
Drug: Umeclidinium/ Vilanterol — Umeclidinium/Vilanterol will be provided as dry white powder for inhalation via a DPI with 30 doses (2 strips with 30 blisters per strip). First strip will contain umeclidinium blended with lactose and magnesium stearate with a unit dose strength of 62.5 mcg per blister and the second strip will contain vilanterol blended with lactose and magnesium stearate with a unit dose strength of 25 mcg per blister
  Arms: UMEC/VI 62.5/25 mcg
Drug: Placebo — Placebo will be provided as dry white powder for inhalation via a DPI with 30 doses (2 strips with 30 blisters per strip) containing lactose
  Arms: Placebo

SUMMARY:
Batefenterol is a novel bifunctional molecule that combines muscarinic antagonism and beta2-agonism in a single molecule. This is a multicenter, randomized, placebo-controlled, double-blind, parallel group study primarily designed to assess the dose response, efficacy and safety of five dose regimens of batefenterol administered via the dry powder inhaler (DPI) once-daily in the morning for 42 days in subjects with COPD. The information obtained from this study will be used to select the minimal, optimally effective and safe dose of batefenterol and also to evaluate the pharmacokinetic profile and established pharmacodynamic (PD) responses of batefenterol. These data will support for future studies with batefenterol in COPD subjects.

The study will consist of a pre-screening visit, screening visit; a run-in period (2 weeks), treatment period of 42 days and a follow-up visit 7 days post-treatment. The total duration of the study for each subject will be approximately 9 weeks. Approximately 460 subjects will be screened in order to randomize approximately 320 subjects, assuming that 280 subjects will complete the study. During treatment period, subjects will be randomized to one of the following treatments delivered via DPI once daily in the morning: Batefenterol 37.5 mcg, 75 mcg, 150 mcg, 300 mcg and 600 mcg, umeclidinium/vilanterol (UMEC/VI) 62.5/25 mcg and placebo. All subjects will receive supplemental albuterol/salbutamol to be used on an as-needed basis (rescue medication) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* Informed Consent: A signed and dated written informed consent prior to study participation
* Age: 40 years of age or older at Visit 1.
* Gender: Male and female subjects are eligible to participate in the study. Female subjects are eligible to participate if not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as:

Pre-menopausal females with one of the following: Documented tubal ligation Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion Hysterectomy Documented Bilateral Oophorectomy Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed below 30 days prior to the first dose of study medication and until at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer after the last dose of study medication and completion of the follow-up visit. This list does not apply to females of reproductive potential with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.

Contraceptive subdermal implant that meets <1 percent (%) rate of failure per year, as stated in the product label Intrauterine device or intrauterine system that meets <1% rate of failure per year, as stated in the product label Oral Contraceptive, either combined or progestogen alone Injectable progestogen Contraceptive vaginal ring Percutaneous contraceptive patches Male partner sterilization with documentation of azoospermia prior to the female subjects entry into the study, and this male is the sole partner for that subject These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society as follows: Chronic obstructive pulmonary disease is a preventable and treatable disease state characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g. 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack-years). Note: pipe and cigar cannot be used to calculate pack-year history.
* Severity of Disease: A post-albuterol/salbutamol FEV1/FVC ratio of <=0.70 and a post-albuterol/salbutamol FEV1 >=30 and <=70% of predicted normal at Visit 1.

Note: Percent predicted will be calculated using the European Respiratory Society Global Lung Function Initiative reference equations.

Exclusion Criteria:

* Asthma: Subjects with a current diagnosis of asthma. (subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Other Respiratory Disorders: Known respiratory disorders other than COPD including but not limited to alpha-1 antitrypsin deficiency, active tuberculosis, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension unrelated to COPD, and interstitial lung disease. Allergic rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Any significant diseases (including uncontrolled hypertension, diabetes and thyroid disease) that in the opinion of the investigator or the study medical monitor would put the safety of the subject at risk through study participation, or which would affect study analyses if the diseases/condition exacerbated during the study.
* Hepatitis: Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening Visit 1 or within 3 months prior to first dose of study treatment. (subjects with positive hepatitis C antibody due to prior resolved disease can be enrolled only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) polymerase chain reaction (PCR) test is obtained).
* Liver Disease: Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Cancer: A current malignancy or previous history of cancer in remission for <5 years prior to Visit 1 (localised basal cell or squamous cell carcinoma of the skin that has been resected is not exclusionary.) Any current or previous history of throat cancer.
* Chest X-Ray: A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Visit 1 if a chest X-ray or CT scan is not available within 6 months prior to Visit 1. For subjects in Germany, if a chest X-ray (or CT scan) is not available in the 6 months prior to Visit 1 the subject will not be eligible for the study.
* Drug Allergy: A history of hypersensitivity or allergy to any beta adrenergic receptor-agonist, sympathomimetic, anticholinergic/anti-muscarinic receptor antagonist, or lactose/milk protein, which in the opinion of the investigator or GlaxoSmithKline (GSK) medical monitor contraindicates study participation.
* Diseases Preventing Use of Anticholinergic: Medical diagnosis of narrow- angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the study investigator would prevent use of an inhaled anticholinergic.
* Poorly controlled COPD: defined as the occurrence of 'acute worsening of COPD that is managed with corticosteroid and/or antibiotics or that requires treatment prescribed by a physician in the 6 weeks prior to Screening (Visit 1), or 'subjects who are hospitalized due to acute worsening of COPD within 12 weeks of Visit 1.
* History of COPD exacerbation: Subjects who have had more than one exacerbation (moderate or severe) within the 12 months prior to Visit 1.
* Pneumonia and lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Visit 1 or subjects hospitalized due to pneumonia within 12 weeks of Visit 1.
* Lung Resection: Lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-lead ECG: An abnormal and clinically significant 12-lead electrocardiogram (ECG). Site investigators will be provided with ECG over-read conducted by a centralized independent cardiologist, to assist in evaluation of subject eligibility. For this study, an abnormal and clinically significant ECG that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to the criteria mentioned in the protocol.
* Screening Labs: Clinically significant abnormal finding from clinical chemistry or hematology tests at Visit 1.
* Medication Prior to Spirometry: Unable to with hold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Excluded Medications: Use of the following medications are not permitted within the defined time intervals prior to Visit 1 and throughout the study: depot corticosteroids (12 weeks), antibiotics (for lower respiratory tract infection) (6 weeks), cytochrome P450 3A4 strong inhibitors and P-glycoprotein inhibitors (4 weeks), systemic, oral or parenteral corticosteroids (2 weeks), inhaled corticosteroids (ICS) or long-acting beta2- agonist (LABA)/ ICS combination products (2 weeks), phosphodiesterase 4 (PDE4) inhibitor (roflumilast) (2 weeks), LABA/ long acting muscarinic receptor antagonist (LAMA) combination (eg vilanterol /umeclidinium bromide) (2 weeks), Once-daily beta2-agonist ( eg Olodaterol and Indacaterol) (10 days), long acting muscarinic antagonists (eg tiotropium, aclidinium, glycopyrronium, umeclidinium) (7 days), theophyllines (48 h), oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) (48 h), oral beta2-agonists long-acting (48 h), short-acting (12 h), inhaled long acting beta2-agonists (LABA, e.g. salmeterol, formoterol, indacaterol) (48 h), inhaled sodium cromoglycate or nedocromil sodium (24 h), inhaled short acting beta2-agonists (4 h), inhaled short-acting anticholinergics (4 h), inhaled short-acting anticholinergic/ short-acting beta2-agonist combination products (4 h), any other investigational medication (30 days or within 5 drug half-lives [whichever is longer]).

The complete list of excluded cytochrome P450 inhibitors and P-glycoprotein inhibitors will be provided in study reference manual (SRM).

Use of study provided albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing.

* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 h a day. As-needed oxygen use (i.e. <=12 h per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g. albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a diary.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (9):
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
- Germany (6):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- South Africa (8):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Meyerspark/ Pretoria
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Thabazimbi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=201012

REFERENCES:
- [Background] Crim C, Watkins ML, Bateman ED, Feldman GJ, Schenkenberger I, Kerwin EM, Crawford C, Pudi K, Ho S, Baidoo C, Castro-Santamaria R. Randomized dose-finding study of batefenterol via dry powder inhaler in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2019 Mar 8;14:615-629. doi: 10.2147/COPD.S190603. eCollection 2019. PMID 30880951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (par.) with an established clinical history of Chronic Obstructive Pulmonary Disease (COPD), were included in this dose-finding study of batefenterol (BAT). Of 585 par. screened, 324 par. were randomized in the study, out of which one par. was randomized in error and was not included in the Intent-to-Treat analysis.
Pre-assignment Details: Pre-bronchodilator and post albuterol/salbutamol spirometry testing were performed at Screening visit. Post-albuterol/salbutamol (Forced expiratory Volume in One Second) FEV1 and FEV1/ (Forced Vital Capacity) FVC values were used to determine subject eligibility. Participants underwent 2 weeks run-in period.
Groups:
- Placebo: Participants received 1 actuation of placebo inhalation powder via Dry Powder Inhaler (DPI) (containing 2 strips) once daily in the morning for 42 days.
- Batefenterol 37.5 µg: Participants received 1 actuation of batefenterol 37.5 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained lactose and second strip contained batefenterol blended with lactose.
- Batefenterol 75 µg: Participants received 1 actuation of batefenterol 75 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained lactose and second strip contained batefenterol blended with lactose.
- Batefenterol 150 µg: Participants received 1 actuation of batefenterol 150 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained lactose and second strip contained batefenterol blended with lactose.
- Batefenterol 300 µg: Participants received 1 actuation of batefenterol 300 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained lactose and second strip contained batefenterol blended with lactose.
- Batefenterol 600 µg: Participants received 1 actuation of batefenterol 600 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained lactose and second strip contained batefenterol blended with lactose.
- UMEC/VI 62.5/25 µg: Participants received 1 actuation of UMEC/VI 62.5/25 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained UMEC blended with lactose and magnesium stearate. Second strip contained VI blended with lactose and magnesium stearate.
Period: Overall Study
Arm/Group | Placebo | Batefenterol 37.5 µg | Batefenterol 75 µg | Batefenterol 150 µg | Batefenterol 300 µg | Batefenterol 600 µg | UMEC/VI 62.5/25 µg
Started | 46 | 46 | 46 | 45 | 47 | 46 | 47
Completed | 44 | 43 | 41 | 40 | 41 | 44 | 47
Not Completed | 2 | 3 | 5 | 5 | 6 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 4 | 0 | 0
Not completed — Par. Reached Stopping Criteria | 1 | 1 | 0 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Par. did not Meet Continuation Criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal Request by GSK | 0 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Batefenterol 37.5 µg | Batefenterol 75 µg | Batefenterol 150 µg | Batefenterol 300 µg | Batefenterol 600 µg | UMEC/VI 62.5/25 µg | Total
Number analyzed (Participants) | 46 | 46 | 46 | 45 | 47 | 46 | 47 | 323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (6.60) | 61.9 (8.16) | 63.0 (7.21) | 63.6 (8.11) | 61.9 (8.70) | 63.7 (7.06) | 62.8 (8.46) | 62.6 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 13 | 26 | 20 | 25 | 21 | 143
  Male | 27 | 27 | 33 | 19 | 27 | 21 | 26 | 180
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6 | 3 | 3 | 2 | 4 | 3 | 2 | 23
  White | 38 | 35 | 40 | 35 | 40 | 38 | 39 | 265
  Multiple Geographic Ancestries | 2 | 8 | 3 | 8 | 3 | 5 | 6 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean FEV1 Over 0 to 6 Hours Post-dose at Day 42
Description: FEV1 is defined as the volume of air that can be forced out in one second after taking a deep breath. Weighted-mean change from Baseline was the weighted-mean FEV1 on Day 42 minus Baseline where Baseline is defined as the average of Day1 pre-dose FEV1 measured at -30 minutes and 0 minutes. The 0-6 hour (Hr.) serial FEV1 was collected at Day 1 (Visit 2) and Day 42 (Visit 6). The weighted-mean was derived by calculating the area under the curve (AUC) of FEV1 over the 6 hour period, and then dividing it by the 6-hour time interval. Batefenterol dose for each individual was compared with placebo or UMEC/VI. The change from Baseline in FEV1 was statistically analyzed using Bayesian Emax modeling of the dose response curve. Intent-to-Treat (ITT) Population comprised of all participants randomized to treatment and who received at least one dose of study medication. Participants with FEV1 values available at Baseline and Day 42 were analyzed.
Time Frame: Baseline and Day 42
Population: ITT Population.
Measure: Mean (Standard Error); unit: Milliliters (mL)
Arm/Group | Placebo | Batefenterol 37.5 µg | Batefenterol 75 µg | Batefenterol 150 µg | Batefenterol 300 µg | Batefenterol 600 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 44 | 42 | 41 | 39 | 41 | 44 | 47
Milliliters (mL) | -9.90 (31.21) | 181.20 (30.85) | 221.68 (21.09) | 251.87 (16.30) | 271.47 (19.49) | 282.94 (24.20) | 275.43 (29.91)
Statistical Analysis 1: Comparison: Placebo vs Batefenterol 37.5 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 191.1, 95% CI 2-sided [101.07 to 284.26] — The 95% Bayesian credible interval for the mean difference between batefenterol 37.5 µg dose and placebo (batefenterol 37.5 µg minus placebo) was estimated
Statistical Analysis 2: Comparison: Placebo vs Batefenterol 75 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 231.6, 95% CI 2-sided [149.31 to 310.02] — The 95% Bayesian credible interval for differences between each individual batefenterol 75 µg dose and placebo was estimated
Statistical Analysis 3: Comparison: Placebo vs Batefenterol 150 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 261.8, 95% CI 2-sided [189.85 to 332.25] — The 95% Bayesian credible interval for differences between each individual batefenterol 150 µg dose and placebo was estimated
Statistical Analysis 4: Comparison: Placebo vs Batefenterol 300 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 281.4, 95% CI 2-sided [212.35 to 351.30] — The 95% Bayesian credible interval for differences between each individual batefenterol 300 µg dose and placebo was estimated
Statistical Analysis 5: Comparison: Placebo vs Batefenterol 600 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 292.8, 95% CI 2-sided [223.02 to 364.42] — The 95% Bayesian credible interval for differences between each individual batefenterol 600 µg dose and placebo was estimated

2. Secondary Outcome: Change From Baseline in Trough FEV1 at Day 42
Description: Trough FEV1 at Day 42 is the mean volume of air that can be forced out in one second after taking a deep breath at the approximately 23 Hrs and 24 Hrs assessments after the last administration of study drug. Batefenterol dose for each individual was compared with placebo or UMEC/VI. Change from Baseline was calculated as trough FEV1 on Day 42 minus baseline, where Baseline is defined as the average of Day1 pre-dose FEV1 measured at -30 minutes and 0 minutes. The Maximum Likelihood Estimation (MLE) method of dose response modeling with Emax modeling without Bayesian priors was used. Participants with FEV1 values available at Baseline and Day 42 after 24 hrs after the last administration of study drug were analyzed.
Time Frame: Baseline and Day 42
Population: ITT Population
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | Batefenterol 37.5 µg | Batefenterol 75 µg | Batefenterol 150 µg | Batefenterol 300 µg | Batefenterol 600 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 44 | 43 | 41 | 40 | 41 | 44 | 47
mL | -35.7 (30.80) | 146.5 (28.30) | 160.8 (15.60) | 168.9 (15.00) | 173.2 (18.20) | 175.4 (20.50) | 209.0 (29.80)
Statistical Analysis 1: Comparison: Placebo vs Batefenterol 37.5 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 182.20, 95% CI 2-sided [99.80 to 264.60] — The 95% confidence interval for the difference between 37.5 µg Batefenterol and Placebo was estimated
Statistical Analysis 2: Comparison: Placebo vs Batefenterol 75 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 196.60, 95% CI 2-sided [128.40 to 264.80] — The 95% confidence interval for the difference between 75 µg Batefenterol and Placebo was estimated
Statistical Analysis 3: Comparison: Placebo vs Batefenterol 150 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 204.60, 95% CI 2-sided [137.20 to 272.10] — The 95% confidence interval for the difference between 150 µg Batefenterol and Placebo was estimated
Statistical Analysis 4: Comparison: Placebo vs Batefenterol 300 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 208.90, 95% CI 2-sided [138.70 to 279.20] — The 95% confidence interval for the difference between 300 µg Batefenterol and Placebo was estimated
Statistical Analysis 5: Comparison: Placebo vs Batefenterol 600 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 211.10, 95% CI 2-sided [138.60 to 283.70] — The 95% confidence interval for the difference between 600 µg Batefenterol and Placebo was estimated

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected from start of study until follow-up contact (Visit7[Visit 6/EW+7days]). Non-serious AEs were collected from start of study treatment (Visit2) until follow-up contact (Visit7[Visit 6/EW+7days]).
Description: AE and SAE analysis was based on ITT Population consisting of all participants randomized to treatment and who received at least one dose of study medication. On-treatment AEs and SAEs were defined as those with onset between treatment start date and treatment stop date +1.
Groups:
- Batefenterol 75 µg: Participants received 1 actuation of batefenterol 75 µg inhalation powder administered via DPI (containing 2 strips) once daily in the morning for 42 days. First strip contained lactose and second strip contained btefenterol blended with lactose.
Arm/Group | Placebo | Batefenterol 37.5 µg | Batefenterol 75 µg | Batefenterol 150 µg | Batefenterol 300 µg | Batefenterol 600 µg | UMEC/VI 62.5/25 µg
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 2/46 | 0/45 | 1/47 | 1/46 | 1/47
Other Adverse Events (participants affected / at risk) | 2/46 | 3/46 | 8/46 | 5/45 | 7/47 | 18/46 | 4/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Batefenterol 37.5 µg (N=46) | Batefenterol 75 µg (N=46) | Batefenterol 150 µg (N=45) | Batefenterol 300 µg (N=47) | Batefenterol 600 µg (N=46) | UMEC/VI 62.5/25 µg (N=47)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Batefenterol 37.5 µg (N=46) | Batefenterol 75 µg (N=46) | Batefenterol 150 µg (N=45) | Batefenterol 300 µg (N=47) | Batefenterol 600 µg (N=46) | UMEC/VI 62.5/25 µg (N=47)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 1 | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 4 | 5 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.